CLINICAL TRIAL: NCT01691118
Title: Fimasartan for Improvement of Diastolic Dysfunction in Hypertensive Patients
Brief Title: A Trial of Fimasartan for Early Diastolic Heart Failure
Acronym: FINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-0229
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension
Keywords: Hypertension; Angiotensin Receptor Blocker; Diastolic Dysfunction
MeSH Terms: conditions — Hypertension | interventions — fimasartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fimasartan (Active Comparator): Fimasartan 60mg qd added on conventional antihypertensive treatment for 10 months.
  Interventions: Drug: Fimasartan; Drug: Antihypertensive treatment
- Placebo (Placebo Comparator): Conventional antihypetensive treatment
  Interventions: Drug: Antihypertensive treatment

INTERVENTIONS:
Drug: Fimasartan
  Arms: Fimasartan
Drug: Antihypertensive treatment

SUMMARY:
Approximately half of hypertensive patients have diastolic dysfunction and diastolic dysfunction is associated with development of congestive heart failure and increased mortality. Although diastolic heart failure associated with hypertension is a clinically significant problem, few clinical trials have been conducted and there is no proven pharmacological therapy to improve outcomes. To the best of the investigators knowledge, there has been no randomized trial to demonstrate that an antihypertensive drug improves diastolic function in hypertensive patients with diastolic dysfunction. The investigators hypothesize that fimasartan added to standard therapy will be superior to placebo in improving diastolic dysfunction in mildly symptomatic patients with hypertension and diastolic dysfunction, and try to examine this hypothesis in a double-blind, randomized comparison study using echocardiography.

DETAILED DESCRIPTION:
Approximately half of hypertensive patients have diastolic dysfunction and diastolic dysfunction is associated with development of congestive heart failure and increased mortality. The Framingham study reported that 51% of patients with HF have a preserved left ventricular (LV) ejection fraction and hypertension is the strongest risk factor for HF with preserved ejection fraction, also termed diastolic heart failure. The rates of death and morbidity in these patients are as high as in patients with HF and a low LV ejection fraction. Hypertensive patients are at increased risk of developing LV hypertrophy and myocardial fibrosis, which cause relaxation abnormality and decreased compliance of LV with a rise in the LV diastolic pressure. Although HF associated with hypertension is a clinically significant problem, few clinical trials have been conducted and there is no proven pharmacological therapy to improve outcomes.

Because the activation of rennin-angiotensin-aldosterone system (RAAS) has been shown to induce LV hypertrophy and myocardial fibrosis, the RAAS may play a central role in the pathogenic process from hypertension to diastolic HF. Inhibitors of RAAS have been considered as a treatment option for these patients, and the angiotensin receptor blockers (ARB) have been of interest because they antagonize the effects of angiotensin II more completely. The largest clinical trial, the Irbesartan in Heart Failure with Preserved Systolic Function (I-PRESERVE), recently reported that treatment with irbesartan did not reduce the risk of death or hospitalization for cardiovascular causes among 4,128 patients who had HF with a preserved LV ejection fraction. The negative result observed in the I-PRESERVE trial may have been the consequence of the following possible factors. First, this trial may have targeted patients in whom the disease process was too advanced for ARBs to be effective. Second, irbesartan may not be an appropriate ARB for a HF trial, because ARBs are not all the same in terms of clinical outcome data in patients with HF. Irbesartan did not have outcome data on reducing HF hospitalization in high-risk hypertensive patients and telmisartan showed no benefits compared to placebo in these patients, although candesartan and valsartan significantly reduced endpoint in placebo-controlled trials. Telmisartan and irbesartan have PPARγ activity and this activity might neutralize the beneficial effects of ARB on HF, because it is well known that PPARγ agonist, rosiglitazone, increases the incidences of HF significantly.

Evaluating the effect of treatments on diastolic dysfunction has been limited by difficulties in non-invasive measure of LV diastolic pressure, but recent advances in echocardiography have made it possible to assess diastolic dysfunction accurately and reproducibly. Thus, additional clinical studies with the other ARBs are needed in hypertensive patients with diastolic dysfunction and assessment of diastolic function by echocardiography will be helpful to determine whether addition of ARB to standard therapy is beneficial to hypertensive patients with diastolic dysfunction. Fimasartan is the first ARB developed in Korea, and was felt to be particularly appropriate for examining the hypothesis that the ARB can improve diastolic dysfunction associated with hypertension, because fimasartan is a potent and well-tolerated ARB. To the best of our knowledge, there has been no randomized trial to demonstrate that an antihypertensive drug improves diastolic function in hypertensive patients with diastolic dysfunction. We hypothesize that fimasartan added to standard therapy will be superior to placebo in improving diastolic dysfunction in mildly symptomatic patients with hypertension and diastolic dysfunction, and try to examine this hypothesis in a double-blind, randomized comparison study using echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Untreated hypertension: systolic BP ≥ 140 or diastolic BP ≥ 90 mmHg or Treated hypertension
* Current heart failure symptoms with NYHA class II
* Evidence of diastolic dysfunction showing any 2 of the following:

E/E' > 10, LV posterior wall thickness > 11 mm, BNP level > 40 pg/mL

Exclusion Criteria:

* Planned cardiac surgery or planned major non-cardiac surgery within the study period
* Stroke or coronary revascularization in the past 6 months
* LV ejection fraction < 50%
* Hypertrophic or restrictive cardiomyopathy, moderate or severe valve disease, constrictive pericarditis
* Atrial fibrillation with a heart rate > 120/min
* Sitting systolic BP < 100 mmHg
* Sitting systolic BP > 160 mmHg or diastolic BP > 95 mmHg despite antihypertensive therapy
* Significant renal disease manifested by serum creatinine > 2.5 mg/dL
* Clinically significant pulmonary disease, coronary artery disease
* A diagnosis of cancer (other than superficial squamous or basal cell skin cancer) in the past 3 years or current treatment for the active cancer
* Female of child-bearing potential who do not use adequate contraception and women who are pregnant or breast-feeding

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in E/E' ratio | 10 months
  Change in the ratio of E velocity (Early mitral inflow velocity) to E' velocity (Early mitral annular velocity) from baseline to 10 months follow-up.

SECONDARY OUTCOMES:
Change in BNP levels | 10 months
  Change in BNP levels from baseline to 10 months follow-up.
Change in left ventricular mass | 10 months
  Change in LV mass from baseline to 10 months follow-up.
Change in left atrial volume | 10 months
  Change in left atrial volume from baseline to 10 months follow-up.
Change in global left ventricular strain | 10 months
  Change in global left ventricular strain from baseline to 10 months follow-up.
Change in functional class | 10 months
  Change in New York Heart Association (NYHA) functional class from baseline to 10 months follow-up.
Change in clinical composite | 10 months
  The clinical composite assessment is based on a change in the NYHA functional class and occurrences of serious adverse events (SAE). Patients with an improvement in NYHA class and without SAE are classified as improved, and those as aggravated if they have SAE during treatment or report worsening of their NYHA class at the endpoint visit.

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hyun Kang, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea